CLINICAL TRIAL: NCT02636218
Title: A Pilot Study of Sub-anesthetic Ketamine Infusion for Neuroprotection After Aneurysmal Subarachnoid Hemorrhage: Effects on White Matter Integrity, Inflammatory Biomarkers and Neurocognitive Outcome
Brief Title: Ketamine Infusion in Neurologic Deficit
Acronym: KIND
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Defence Research and Development Canada (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KTM-3007
Record Dates: First submitted 2015-12-08; First posted 2015-12-21 (Estimated); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Ketamine
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.9% NaCl control (Active Comparator): Normal saline
  Interventions: Drug: 0.9% NaCl
- Ketamine (Experimental): Anesthetic
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — 500 ml of ketamine (0.2 mg/ml) infused at 5 ug/kg/min for 4 hours.
  Other Names: Ketamine HCl
  Arms: Ketamine
Drug: 0.9% NaCl — 500 ml of 0.9% NaCl infused at 5 ug/kg/min for 4 hours.
  Other Names: NS
  Arms: 0.9% NaCl control

SUMMARY:
Subarachnoid hemorrhage (SAH) or bleeding in the brain as a result of ruptured aneurysm is a devastating type of stroke. Many patients who undergo emergent neurosurgery to repair the aneurysm and remove the bleeding suffer from complications in their subsequent hospital stay, the most frequent and morbid of which is delayed cerebral ischemia (DCI) or small strokes resulting from impaired blood flow to certain vital brain centers. This occurs because of changes to the brain's blood vessels that occur after the bleed. The arteries can become narrow (spasm) or small clots can form within the vasculature that disrupts normal blood flow. Patients are left with profound neurologic deficits from these secondary complications.

Anesthesiologists, neurosurgeons, and intensivists are in need of a way to protect the brain during this vulnerable period following aneurysm repair. One drug that may provide such protection is ketamine, a compound frequently used in operating rooms and intensive care units to provide anesthesia and analgesia. Ketamine works by blocking glutamate receptor ion channels that play a pivotal role in promoting brain cell death during strokes by flooding the brain with too much calcium and dangerous chemicals. This project is designed to test the efficacy of ketamine in protecting the brain following aneurysm repair by using a controlled infusion of the drug in the intensive care unit (ICU) when patients return from their operation.

DETAILED DESCRIPTION:
Aneurysmal subarachnoid hemorrhage (aSAH) is a devastating type of stroke, with significant long-term morbidity for patients who survive the initial bleed. The most frequent and morbid complication is delayed cerebral ischemia (DCI) resulting from angiographic vasospasm of the arteries of the circle of Willis. At present, there is no protective therapy aimed at neuronal preservation during this period of ischemia. The standard medical care is primarily to maintain intravascular volume status to improve cerebral perfusion during arterial narrowing, or calcium channel blockers for smooth muscle relaxation on the arterial wall. Experimental and clinical data suggest a primary mechanism of neuronal injury during ischemia is excitotoxicity, glutamate-induced cell death resulting from overstimulation of ionotropic N-methyl-D-aspartate (NMDA) receptors and resultant excessive calcium influx. Ketamine is a dissociative anesthetic with a mechanism of action of non-competitive antagonism of the NMDA receptor, routinely used in operating rooms and intensive care units as an analgesic and anesthetic. In addition to its anesthetic properties, ketamine is also an anti-inflammatory agent and a sympathomimetic, maintaining sedation without the adverse effects of hemodynamic instability. Identification of a neuroprotective entity for DCI following SAH would vastly improve the quality of life and shorten hospital stay for patients with a ruptured intracerebral aneurysm. It is critical to identify such agents so that patients survive their injury, spend shorter time in the ICU, and can return to work and maintain relationships.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 80 years old.
2. World Federation of Neurological Surgeons (WFNS) grade 2 to 4, obtained after resuscitation and prior to dosing.
3. SAH on admission cranial computed tomography (CT) scan (diffuse clot present in both hemispheres, thin or thick [>4 mm], or local thick SAH (>4 mm).
4. Ruptured saccular aneurysm, confirmed by catheter angiography (CA) or CT angiography (CTA) and treated by neurosurgical clipping or endovascular coiling.
5. External ventricular drain placed as part of routine care.
6. Able to be dosed within 4 hours of new neurologic deficit.
7. Historical modified Rankin score of 0 or 1.
8. Hemodynamically stable after resuscitation (systolic blood pressure > 100 mm Hg)
9. Haemoglobin >85 g/L, platelets >125,000 cells/mm3
10. Informed consent.
11. New neurologic deficits that were not present previously, identified by 1) a decrease of 2 points on the modified Glasgow coma scale (mGCS) or 2) an increase in 2 points on the National Institute of Health Stroke Scale (NIHSS). i.e., a CODE VASOSPASM initiated in the ICU.

Exclusion Criteria:

1. Subarachnoid hemorrhage due to causes other than a saccular aneurysm (e.g., trauma or rupture of fusiform or infective aneurysm).
2. WFNS Grade 1 or 5 assessed after the completion of aneurysm repair.
3. Increased intracranial pressure (ICP) >30 mm Hg in sedated patients lasting >4 hours anytime since admission.
4. Intraventricular or intracerebral hemorrhage in absence of SAH or with only local, thin SAH.
5. Angiographic vasospasm prior to aneurysm repair procedure, as documented by catheter angiogram or CT angiogram.
6. Major complication during aneurysm repair such as, but not limited to, massive intraoperative hemorrhage, brain swelling, arterial occlusion, or inability to secure the ruptured aneurysm.
7. Aneurysm repair requiring flow diverting stent or stent-assisted coiling and dual antiplatelet therapy.
8. Hemodynamically unstable prior to administration of study drug (i.e., SBP <90 mm Hg, requiring >6 L colloid or crystalloid fluid resuscitation).
9. Cardiopulmonary resuscitation was required following SAH.
10. Female patients with positive pregnancy test (blood or urine) at screening.
11. History within the past 6 months and/or physical finding on admission of decompensated heart failure (New York Heart Association [NYHA] Class III and IV or heart failure requiring hospitalization).
12. Acute myocardial infarction within 3 months prior to the administration of the study drug.
13. Symptoms or electrocardiogram (ECG)-based signs of acute myocardial infarction or unstable angina pectoris on admission.
14. Electrocardiogram evidence and/or physical findings compatible with second or third degree heart block or of cardiac arrhythmia associated with hemodynamic instability.
15. Echocardiogram, if performed as part of standard-of-care before treatment, revealing a left ventricular ejection fraction (LVEF) <40%.
16. Severe or unstable concomitant condition or disease (e.g., known significant neurologic deficit, cancer, hematologic, or coronary disease), or chronic condition (e.g., psychiatric disorder) that, in the opinion of the Investigator, may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results.
17. Patients who have received an investigational product or participated in another interventional clinical study within 30 days prior to randomization.
18. Kidney disease as defined by plasma creatinine ≥2.5 mg/dl (221 umol/l); liver disease as defined by total bilirubin >3 mg/dl (51.3 mmol/l); and/or known diagnosis or clinical suspicion of liver cirrhosis.
19. Known hypersensitivity or contraindication to ketamine per product monograph.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Changes in physiologic parameters as specified below | During infusion and 1 hour post-infusion
  Temperature, heart rate (HR), mean arterial pressure (MAP), intracranial pressure (ICP), central venous pressure (CVP) if available, peak airway pressure (PAP) if available, end-tidal carbon dioxide (ETCO2) will be evaluated during infusion. Collected measurement data will be analyzed based on the occurrence of adverse events such as increase in ICP by more than 3 mmHg, increase in HR by more than 30 bpm, increase in partial pressure of CO2 (pCO2) by more than 20 mmHg, increase in lactate by more than 0.5, drop in pH by more than 0.2, increase in systolic blood pressure (SBP0 to over 200 mmHg, or any other unforeseen event that is deemed to be related to the drug treatment with adverse effects on the patient.

SECONDARY OUTCOMES:
Biologic samples | Day 1-2 post-infusion
  Blood and cerebrospinal fluid (CSF) samples will be collected and analyzed for biomarker levels which would indicate extent of neuronal injury.
Neurocognitive test Montreal Cognitive Assessment Scale (MoCA) | Day 30 or Day 60 post-DCI
  Neurocognitive function will be assessed using the MoCA to determine preliminary effects of ketamine on neurocognitive outcome.
Neurocognitive test modified Rankin Scale (mRS) | Day 30 or Day 60 post-DCI
  Neurocognitive function will be assessed using the mRS determine preliminary effects of ketamine on neurocognitive outcome.
Brain imaging using Magnetic Resonance Imaging (MRI) | Day 30 or Day 60 post-DCI
  Structural and functional brain imaging will be conducted using Tesla MRI system to assess white matter integrity.
Hospital anxiety and depression score | Day 30 or Day 60 post-DCI
  Assessments for neuro-cognitive outcomes and correlation with MRI findings
EQ-5D-5L | Day 30 or Day 60 post-DCI
  Neurocognitive outcome assessment and correlation with MRI results
Trail making test | Day 30 or Day 60 post-DCI
  Neurocognitive outcome assessment and correlation with MRI results
Verbal fluency tests | Day 30 or Day 60 post-DCI
  Neurocognitive outcome assessment and correlation with MRI results

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Baker, MD, FRCPC, Principal Investigator — Unity Health Toronto
Locations (1):
- St Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Etminan N, Vergouwen MD, Ilodigwe D, Macdonald RL. Effect of pharmaceutical treatment on vasospasm, delayed cerebral ischemia, and clinical outcome in patients with aneurysmal subarachnoid hemorrhage: a systematic review and meta-analysis. J Cereb Blood Flow Metab. 2011 Jun;31(6):1443-51. doi: 10.1038/jcbfm.2011.7. Epub 2011 Feb 2. PMID 21285966
- [Background] Nilsson OG, Saveland H, Boris-Moller F, Brandt L, Wieloch T. Increased levels of glutamate in patients with subarachnoid haemorrhage as measured by intracerebral microdialysis. Acta Neurochir Suppl. 1996;67:45-7. doi: 10.1007/978-3-7091-6894-3_10. PMID 8870801
- [Background] Beal MF. Mechanisms of excitotoxicity in neurologic diseases. FASEB J. 1992 Dec;6(15):3338-44. PMID 1464368
- [Background] Forder JP, Tymianski M. Postsynaptic mechanisms of excitotoxicity: Involvement of postsynaptic density proteins, radicals, and oxidant molecules. Neuroscience. 2009 Jan 12;158(1):293-300. doi: 10.1016/j.neuroscience.2008.10.021. Epub 2008 Nov 1. PMID 19041375